CLINICAL TRIAL: NCT06099964
Title: Brief Mindfulness Intervention for a Heterogenous Mix of Orthopedic Patients
Brief Title: Brief Mindfulness Intervention for Orthopedic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB_00085446 2
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Coping Information (Active Comparator): Participants will be randomized to listen to a 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Interventions: Behavioral: Pain Coping Information
- Mindful Pain Management (Experimental): Participants will be randomized to listen to a 4-minute audio recording consisting of a 1-minute introduction to mindfulness followed by a 1-minute and 30-second mindful breathing practice and a 1-minute and 30-second mindfulness of pain practice.
  Interventions: Behavioral: Mindful Pain Management

INTERVENTIONS:
Behavioral: Pain Coping Information — A 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Arms: Pain Coping Information
Behavioral: Mindful Pain Management — A 4-minute audio recording consisting of a 1-minute introduction to mindfulness followed by a 1-minute and 30-second mindful breathing practice and a 1-minute and 30-second mindfulness of pain practice.
  Arms: Mindful Pain Management

SUMMARY:
This is a single-site, two-arm, parallel-group randomized clinical trial (RCT). The clinical effects of a 4-minute audio-recorded mindfulness intervention for orthopedic patients will be investigated relative to a 4-minute audio-recoding about pain psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Seeking foot or ankle treatment at the Tallahassee Orthopedic Center

Exclusion Criteria:

* • Cognitive impairment preventing completion of study procedures.

  * Current cancer diagnosis,
  * Other unstable illness judged by medical staff to interfere with study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Anxiety Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no anxiety and 10 representing severe anxiety.
Change in Depression Numeric Rating Scale | Immediately before to after 4-minute audio recording]
  Single Likert scale item ranging from 0-10, with 0 indicating no depression and 10 indicating severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
All data is aggregated and anonymous.

REFERENCES:
- [Derived] Hanley AW, Wilson Zingg R, Smith B, Zappa M, White S, Davis A, Worts PR, Culjat C, Martorella G. Mindfulness in the Clinic Waiting Room May Decrease Pain: Results from Three Pilot Randomized Controlled Trials. J Integr Complement Med. 2024 Nov;30(11):1082-1091. doi: 10.1089/jicm.2024.0020. Epub 2024 May 17. PMID 38757714